CLINICAL TRIAL: NCT02566109
Title: Community Hospital Identification of High CV Risk Patients During Cancer Treatment (CHI)
Brief Title: Community Hospital Identification of High CV Risk Patients During Cancer Treatment
Acronym: CHI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Issues
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00032416; WF-01115 (Other: NCI)
Record Dates: First submitted 2015-09-28; First posted 2015-10-02 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fast MRI (Other): All patients who agree to participate in this study will have a 10 minute fast MRI scan and Baseline and 6 month time periods. The fast MRI will be used to determine if cardiovascular injury can be detected early while patients are receiving chemotherapy treatment.
  Interventions: Diagnostic Test: Fast MRI

INTERVENTIONS:
Diagnostic Test: Fast MRI — The fast MRI is a 10 minute MRI scan that will be used to determine if cardiovascular injury can be detected early while patients are receiving chemotherapy treatment.

SUMMARY:
The overall of this proposal is to test in community hospitals the utility of a 10-min magnetic resonance imaging (MRI) scan protocol combined with proprietary image analysis algorithms for detecting early cardiovascular (CV) injury during receipt of chemotherapy for breast cancer (BrC) and lymphoma. This technology provides health-care delivery systems with a time-efficient method to identify those at risk of a future CV event so that prevention can be implemented to prolong survival and reduce morbidity in cancer survivors.

DETAILED DESCRIPTION:
While recent research indicates that conventional MRI, advanced echocardiography (global longitudinal strain and 3D) and serum biomarkers can detect CV injury early after receipt of Chemotherapy, these methods require lengthy and difficult examinations that are not routinely executed in community hospitals where the majority of patients with BrC & lymphoma are treated. Yet, 1-month deteriorations in traditional 45-min MRI measures are known to forecast 6-month subclinical deteriorations in left ventricular ejection fraction (LVEF) that are associated with CV events. At the same time, new observational data indicate therapy with HMG-CoA reductase inhibitors/statins administered early during receipt of Chemotherapy may prevent subsequent cardiac dysfunction and CV events. Our MRI fast scanning techniques remedy these community hospital implementation obstacles.

In this proposal, the investigators propose to test the utility of these fast scans within an existing funded randomized clinical trial R01HL118740 of generic atorvastatin that is researching methods to prevent cardiotoxicity in patients treated with Chemotherapy for BrC and lymphoma (taking advantage of significant existing clinical trial resources). This study allows us to address our over-arching goal: to determine the optimal implementation (alone or in combination with other tests) of our proprietary MRI processes for forecasting CV injury in patients treated with Chemotherapy in community hospitals through performance of a Phase II comparative effectiveness study within an ongoing clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Stage I-III breast cancer (including inflammatory and newly diagnosed recurrent breast cancer) or lymphoma with a > 2 year life expectancy
* Scheduled to receive chemotherapy with an Anthracycline (doxorubicin or epirubicin)
* = or > 21 years of age
* Prior cancers allowed if no evidence of disease
* ECOG 0 or 1
* Enrollment in NCI Protocol #: WF 98213. Patients must receive Fast MRI and 3D ECHO along with Baseline (98213) MRI prior to first chemotherapy treatment.

Exclusion Criteria:

* Patients with ferromagnetic cerebral aneurysm clips or other intraorbital/intracranial metal; pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices.
* Most breast tissue expanders are not allowed. (If uncertain, inform the MRI tech to confirm eligibility status.)
* Unable to provide informed consent
* Symptomatic Claustrophobia
* Pregnant or breasting feeding. Due to unknown risks and potential harm to the unborn fetus a negative serum pregnancy test within 10 days prior to registration is required in patients with child-bearing potential. For this reason patients of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence (not having sex), oral contraceptives, intrauterine device (IUD), DeProvera, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). An acceptable, although less reliable method involves the careful use of condoms and spermicidal foam or gel and/or cervical cap or sponge prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hundley, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fast MRI
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Same as total enrolled.
Arm/Group | Fast MRI
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: percentage of fluid expelled] — Population: 1 patient did not receive baseline MRI
  percentage of fluid expelled
    number analyzed (Participants) | 5
    (all) | 61.51 (5.45)
End Diastolic Volume (EDV) - Magnetic Resonance Imaging (MRI) [Mean (Standard Deviation); unit: mL] — Population: 1 patient did not receive baseline MRI
  mL
    number analyzed (Participants) | 5
    (all) | 134.90 (41.70)
End Systolic Volume (ESV) - Magnetic Resonance Imaging (MRI) [Mean (Standard Deviation); unit: mL] — Population: 1 patient did not receive baseline MRI
  mL
    number analyzed (Participants) | 5
    (all) | 52.23 (18.91)
Pulse Wave Velocity (PWV) - Magnetic Resonance Imaging (MRI) [Mean (Standard Deviation); unit: meters/sec] — Population: 1 patient did not receive baseline MRI
  meters/sec
    number analyzed (Participants) | 5
    (all) | 4.74 (1.75)
Left Ventricular Ejection Fraction (LVEF) - Echocardiogram (ECHO) [Mean (Standard Deviation); unit: percentage of fluid expelled] | 54.17 (7.03)
End Diastolic Volume (EDV) - Echocardiogram (ECHO) [Mean (Standard Deviation); unit: mL] | 100.08 (24.20)
End Systolic Volume (ESV) - Echocardiogram (ECHO) [Mean (Standard Deviation); unit: mL] | 44.90 (9.16)

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF) at Baseline, 2 Month Using Fast MRI, and 6 Months
Description: To compare baseline, 2-month (using Fast MRI), and 6 month measures in left ventricular (LV) ejection fraction
Time Frame: Baseline, 2 months, and 6 months
Population: Only 5 received MRI at baseline, 4 at 2 months using Fast MRI, and 3 at 6 months.
Measure: Mean (Standard Deviation); unit: percentage of fluid ejected
Arm/Group | Fast MRI
Number analyzed (Participants) | 5
percentage of fluid ejected
  2 months FAST MRI: number analyzed (Participants) | 4
  2 months FAST MRI | 56.67 (4.71)
  6 months: number analyzed (Participants) | 3
  6 months | 58.69 (3.28)
Statistical Analysis 1: Comparison: Fast MRI; Correlation between baseline and 2 months; Test type: Other — Estimation of Pearson correlation; p = 0.6102, Pearson Correlation Coefficient; Pearson Correlation Coefficient = -0.57472
Statistical Analysis 2: Comparison: Fast MRI; Correlation between baseline and 6 months; Test type: Other — Correlation; p = 0.8343, Peason Correlation Coefficient; Pearson Correlation Coefficient = 0.25733

2. Primary Outcome: End Diastolic Volume (EDV) at Baseline, 2 Month, and 6 Months
Description: To compare baseline, 2-month (using Fast MRI), and 6 month measures in end Diastolic Volume (EDV)
Time Frame: Baseline, 2 months, and 6 months
Population: Only 5 received MRI at baseline, 4 at 2 months using Fast MRI, and 3 at 6 months.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Fast MRI
Number analyzed (Participants) | 5
mL
  2 months FAST MRI: number analyzed (Participants) | 4
  2 months FAST MRI | 126.07 (32.36)
  6 months: number analyzed (Participants) | 3
  6 months | 130.20 (44.52)
Statistical Analysis 1: Comparison: Fast MRI; Correlation between baseline and 2 months; Test type: Other — Pearson Correlation Coefficient; p = 0.9395, Pearson Correlation Coefficient; Pearson Correlation Coefficient = -0.09487
Statistical Analysis 2: Comparison: Fast MRI; Correlation between baseline and 6 months; Test type: Other — Pearson Correlation Coefficient; p = 0.1486, Pearson Correlation Coefficient; Pearson Correlation Coefficient = 0.97287

3. Primary Outcome: End Systolic Volume (ESV) at Baseline, 2 Month, and 6 Months
Description: To compare baseline, 2-month (using Fast MRI), and 6 month measures in end Systolic Volume (ESV)
Time Frame: Baseline, 2 months, and 6 months
Population: Only 5 received MRI at baseline, 4 at 2 months using Fast MRI, and 3 at 6 months.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Fast MRI
Number analyzed (Participants) | 5
mL
  2 months FAST MRI: number analyzed (Participants) | 4
  2 months FAST MRI | 54.72 (14.52)
  6 months: number analyzed (Participants) | 3
  6 months | 54.73 (23.11)
Statistical Analysis 1: Comparison: Fast MRI; Correlation between baseline and 2 months; Test type: Other — Pearson Correlation Coefficient; p = 0.9341, Pearson Correlation Coefficient; Pearson Correlation Coefficient = 0.10327
Statistical Analysis 2: Comparison: Fast MRI; Correlation between baseline and 6 months; Test type: Other — Pearson Correlation Coefficient; p = 0.0497, Pearson Correlation Coefficient; Pearson Correlation Coefficient = 0.99696

4. Primary Outcome: Pulse Wave Velocity (PWV) at Baseline and 6 Months
Description: To compare baseline and 6 month measures in pulse wave velocity (PWV)
Time Frame: Baseline and 6 months
Population: Only 5 received MRI at baseline and 3 at 6 months.
Measure: Mean (Standard Deviation); unit: Meters/sec
Arm/Group | Fast MRI
Number analyzed (Participants) | 5
Meters/sec
  Baseline | 4.74 (1.75)
  6 months: number analyzed (Participants) | 3
  6 months | 4.07 (1.70)
Statistical Analysis 1: Comparison: Fast MRI; Test type: Other — Pearson Correlation Coefficient; p = 0.1129, Pearson Correlation Coefficient; Pearson Correlation Coefficient = 0.98432

5. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF): Comparison of Magnetic Resonance Imaging (MRI) With Echocardiogram (ECHO) at Baseline
Description: To compare Magnetic Resonance Imaging (MRI) metric of Left Ventricular Ejection Fraction (LVEF) with Echocardiogram (ECHO) at baseline
Time Frame: Baseline
Population: All 6 participants that received both an ECHO. Only 5 had an MRI at baseline
Measure: Mean (Standard Deviation); unit: percentage of fluid expelled
Arm/Group | Fast MRI
Number analyzed (Participants) | 6
percentage of fluid expelled
  LVEF Echo | 54.17 (7.03)
  LVEF MRI: number analyzed (Participants) | 5
  LVEF MRI | 61.51 (5.45)

6. Secondary Outcome: End Diastolic Volume (EDV): Compare Magnetic Resonance Imaging (MRI) With Echocardiogram (ECHO) at Baseline
Description: To compare magnetic resonance imaging (MRI) metric of End Diastolic Volume (EDV) with echocardiogram (ECHO) at baseline
Time Frame: Baseline
Population: All 6 participants that received both an ECHO. Only 5 had an MRI at baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Fast MRI
Number analyzed (Participants) | 6
mL
  EDV Echo | 100.08 (24.20)
  EDV MRI: number analyzed (Participants) | 5
  EDV MRI | 134.90 (41.70)

7. Secondary Outcome: End Systolic Volume (ESV): Compare Magnetic Resonance Imaging (MRI) With Echocardiogram (ECHO) at Baseline
Description: To compare magnetic resonance imaging (MRI) metric of End Systolic Volume (ESV) with echocardiogram (ECHO) at baseline
Time Frame: Baseline
Population: All 6 participants that received both an ECHO. Only 5 had an MRI at baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Fast MRI
Number analyzed (Participants) | 6
mL
  ESV Echo | 44.90 (9.16)
  ESV MRI: number analyzed (Participants) | 5
  ESV MRI | 52.23 (18.91)

8. Other Pre Specified Outcome: Exploratory Algorithmic Modeling
Description: To use exploratory algorithmic modeling to obtain optimal strategies for determining the combination of metrics (10-min MR, ECHO, serum biomarkers) at 2-months that predict the 6-month post Chemotherapy deteriorations in cardiovascular function.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of signed informed consent to 30 days post study completion for each participant. Study completion was approximately 6 months.
Description: Grades 1, 2, and 3 expected (solicited) and unexpected (unsolicited) adverse events (AE)s that meet the above definition for an AE and are only definitely related, possibly related or probably related to this study intervention should be reported using the Toxicity Assessment Sheet. Hospitalizations that are scheduled for routine treatments and procedures unrelated to study intervention do not need to be reported. All toxicities are graded using CTCAE v4.03.
Arm/Group | Fast MRI
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast MRI (N=6)
Febrile neutropenia (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subject analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT02566109/Prot_SAP_000.pdf